CLINICAL TRIAL: NCT04486352
Title: A Phase IB/II Multi-Cohort Study of Targeted Agents and/or Immunotherapy With Atezolizumab for Patients With Recurrent or Persistent Endometrial Cancer
Brief Title: A Study of Targeted Agents for Patients With Recurrent or Persistent Endometrial Cancer
Acronym: EndoMAP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Genentech, Inc. (Industry); Foundation Medicine (Industry); Pfizer (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFT-50
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — atezolizumab; Bevacizumab; ipatasertib; talazoparib; Ado-Trastuzumab Emtansine; Tiragolumab; inavolisib; Letrozole; giredestrant; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Atezolizumab and Bevacizumab Cohort - Closed to Accrual (Experimental): Following the submission of tumor tissue for the FoundationOne® companion diagnostic (F1CDx) test, participants with no specified gene signatures will be enrolled in this cohort. Twenty participants will be enrolled. Once twenty participants are enrolled, the cohort will be closed to further enrollment. Participants in this study cohort will commence treatment as specified on Day 1 of each cycle.
  Interventions: Drug: Atezolizumab - 28 Day Cycle; Drug: Bevacizumab
- Atezolizumab and Ipatasertib Cohort - Closed to Accrual (Experimental): Following the submission of tumor tissue for the FoundationOne® companion diagnostic (F1CDx) test, participants with PIK3CA/AKT1/PTEN-altered tumors will be enrolled in this cohort. Twenty participants will be enrolled. Once twenty participants are enrolled, the cohort will be closed to further enrollment. Participants in this study cohort will commence treatment as specified on Day 1 of each cycle.
  Interventions: Drug: Atezolizumab - 28 Day Cycle; Drug: Ipatasertib
- Atezolizumab and Talazoparib Cohort (Experimental): Following the submission of tumor tissue for the FoundationOne® companion diagnostic (F1CDx) test, participants with tumors that have a ≥16%genomic loss of heterozygosity (LOH) will be assigned to this cohort. Twenty participants will be enrolled. Once twenty participants are enrolled, the cohort will be closed to further enrollment. Participants in this study cohort will commence treatment as specified on Day 1 of each cycle.
  Interventions: Drug: Atezolizumab - 28 Day Cycle; Drug: Talazoparib
- Atezolizumab and Trastuzumab emtansine (TDM-1) Cohort - Closed to Accrual (Experimental): Following the submission of tumor tissue for the FoundationOne® companion diagnostic (F1CDx) test, participants with tumors that with an amplification of ERBB2/HER2 will be assigned to this cohort. Twenty participants will be enrolled. Once twenty participants are enrolled, the cohort will be closed to further enrollment. Participants in this study cohort will commence treatment as specified on Day 1 of each cycle.
  Interventions: Drug: Trastuzumab emtansine; Drug: Atezolizumab - 21 Day Cycle
- Atezolizumab and Tiragolumab Cohort - Closed to Accrual (Experimental): Following the submission of tumor tissue for the FoundationOne® companion diagnostic (F1CDx) test, participants with tumor type MSI-H and/or tTMB >=10 mut/mb will be assigned to this cohort. Twenty participants will be enrolled initially. Once twenty participants are enrolled, the cohort may be expanded if a positive signal is shown. Participants in this study cohort will commence treatment as specified on Day 1 of each cycle.
  Interventions: Drug: Atezolizumab - 28 Day Cycle; Drug: Tiragolumab
- Inavolisib and Letrozole Cohort (Experimental): Following the submission of tumor tissue for the FoundationOne® companion diagnostic (F1CDx) test, participants with tumors that with PIK3CA activating mutations in the absence of PTEN loss-of-function alterations or AKT1 activating mutations will be assigned to this cohort. Twenty-four participants will be enrolled. Once twenty-four participants are enrolled, the cohort will be closed to further enrollment. Participants in this study cohort will commence treatment as specified on Day 1 of each cycle.
  Interventions: Drug: Inavolisib; Drug: Letrozole
- Giredestrant and Abemaciclib (Experimental): Following the submission of tumor tissue for the FoundationOne® companion diagnostic (F1CDx) test, participants with tumors that are RB1 intact with a local grade 1-2 estrogne receptor positive (ER+) are assigned to this cohort. Twenty-four participants will be enrolled. Once twenty-four participants are enrolled, the cohort will be closed to further enrollment. Participants in this study cohort will commence treatment as specified on Day 1 of each cycle.
  Interventions: Drug: Giredestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Atezolizumab - 28 Day Cycle — Atezolizumab will be given to participants intravenously at a dosage of 1680 mg on day 1 of each 28-day cycle.
  Other Names: Tecentriq; L01XC32
  Arms: Atezolizumab and Bevacizumab Cohort - Closed to Accrual; Atezolizumab and Ipatasertib Cohort - Closed to Accrual; Atezolizumab and Talazoparib Cohort; Atezolizumab and Tiragolumab Cohort - Closed to Accrual
Drug: Bevacizumab — Bevacizumab will be given to participants intravenously at a dosage of 10mg per participant kilogram every 2 weeks of the 28-day cycle.
  Other Names: Avastin; L01XC07
  Arms: Atezolizumab and Bevacizumab Cohort - Closed to Accrual
Drug: Ipatasertib — Ipatasertib will be given as an orally at a dosage of 400 mg once daily for 21 days of each 28-day cycle.
  Other Names: RG7440; GDC-0068
  Arms: Atezolizumab and Ipatasertib Cohort - Closed to Accrual
Drug: Talazoparib — Talazoparib will be given in an orally at a dosage of 1 mg once daily for each day of the 28-day cycle.
  Other Names: Talzenna; L01XX60
  Arms: Atezolizumab and Talazoparib Cohort
Drug: Trastuzumab emtansine — Trastuzumab emtansine be given to participants intravenously at a dosage of 3.6 mg per participant kilogram, on day 1 of each 21-day cycle.
  Other Names: T-DM1; Kadcyla
  Arms: Atezolizumab and Trastuzumab emtansine (TDM-1) Cohort - Closed to Accrual
Drug: Tiragolumab — Tiragolumab will be given to participants intravenously at a dosage of 840 mg on day 1 of each 28-day cycle.
  Arms: Atezolizumab and Tiragolumab Cohort - Closed to Accrual
Drug: Atezolizumab - 21 Day Cycle — Atezolizumab will be given to participants intravenously at a dosage of 1200 mg on day 1 of each 21-day cycle.
  Other Names: Tecentriq; L01XC32
  Arms: Atezolizumab and Trastuzumab emtansine (TDM-1) Cohort - Closed to Accrual
Drug: Inavolisib — Inavolisib will be given in an orally at a dosage of 9 mg once daily for each day of the 28-day cycle.
  Other Names: GDC-0077
  Arms: Inavolisib and Letrozole Cohort
Drug: Letrozole — Letrozole will be given orally at a dosage of 2.5 mg once daily for each day of the 28-day cycle.
  Other Names: Femara
  Arms: Inavolisib and Letrozole Cohort
Drug: Giredestrant — Giredestrant will be given orally at a dosage of 30 mg once daily for each day of the 28-day cycle.
  Other Names: GDC-9545
  Arms: Giredestrant and Abemaciclib
Drug: Abemaciclib — Giredestrant will be given orally at a dosage of 150 mg twice daily for each day of the 28-day cycle.
  Other Names: Verzenio
  Arms: Giredestrant and Abemaciclib

SUMMARY:
This is a Phase IB/II multi-cohort study designed to evaluate the efficacy and safety of targeted agents with or without cancer immune checkpoint therapy with atezolizumab in participant with recurrent and/or persistent endometrial cancer. The main protocol provides a platform for genomic screening with homogeneous basic eligibility criteria in order to direct study participants into biomarker-matched study cohorts consisting of testing targeted agents.

DETAILED DESCRIPTION:
This is a Phase IB/II multi-cohort study designed to evaluate the efficacy and safety of targeted agents with or without cancer immune checkpoint therapy with atezolizumab in participants with recurrent and/or persistent endometrial cancer.

This biomarker-driven study provides a platform whereby participants with persistent/recurrent endometrial cancer will be placed into study cohorts evaluating targeted agents selected on the basis of the tumor's specific genomic profile. Prospective participants with persistent and/or recurrent endometrial cancer will be prescreened within 60 days of treatment assignment to have a tumor tissue sample submitted for next-generation sequencing (NGS) using FoundationOne® companion diagnostic (CDx) testing prior to entering screening. If a participant has FoundationOne® CDx testing within five years of enrollment, the previous tumor tissue may be re-analyzed for use in the study. Non-FMI NGS testing may be submitted if approved.

Depending on the cohort assignment per the tumor's biomarker profile, participants will be assigned to the AFT-50A Protocol (atezolizumab+targeted agent) or the AFT-50B Protocol (non-atezolizumab targeted agents). The current study cohorts are as follows:

AFT-50A Cohorts

* Atezolizumab + Bevacizumab doublet - Closed to Accrual
* Atezolizumab + Ipatasertib doublet - Closed to Accrual
* Atezolizumab + Talazoparib doublet
* Atezolizumab + Trastuzumab emtansine (TDM-1) doublet - Closed to Accrual
* Atezolizumab + Tiragolumab doublet - Closed to Accrual

AFT-50B Cohorts

* Inavolisib + Letrozole doublet
* Giredestrant + Abemaciclib doublet

It is anticipated that approximately 20 participants will be enrolled in each study cohort in AFT-50A and 24 participants in each study cohort in AFT-50B, unless otherwise specified for a given cohort due to statistical considerations. Each study cohort will open/close independently of other study cohorts. Once a study cohort reaches the prespecified number of participants, it will be closed to further enrollment, unless an expansion phase is planned.

The study is structured to allow for additional cohorts to be added as the study progresses. These additional study cohorts may be proposed by investigators, but requires approval by the Steering Committee in order to be added to the protocol.

ELIGIBILITY:
Key Inclusion Criteria:

* Recurrent or persistent endometrial carcinoma which has progressed or recurred after at least 1, but no more than 2, prior lines of therapy. Prior hormonal therapies (e.g., tamoxifen, aromatase inhibitors) will not count toward the prior regimen limit. Chemotherapy given in conjunction with radiotherapy as a radiosensitizer will be counted as a systemic therapeutic regimen.
* Measurable disease per RECIST 1.1
* Availability of a representative tumor specimen that is suitable for determination of biomarker status via central testing (F1CDx) OR If a patient has a prior F1CDx report from 1 September 2019 or later, those NGS results can be used to determine biomarker status as long as the tumor tissue used in the report was obtained within 5 years prior to prescreening and appropriate signed consent is obtained from the patient.
* Life expectancy > 12 weeks
* Recovery from effects of recent radiotherapy, surgery, or chemotherapy

Key Exclusion Criteria:

* Endometrial tumors with the following histologies: squamous carcinomas, sarcomas
* Other invasive malignancies within the last 5 years, except for non-melanoma skin cancer with no evidence of disease within the past 5 years AND localized breast cancer with previous adjuvant chemotherapy treatment for breast cancer completed > 5 years ago
* Synchronous primary invasive ovarian or cervical cancer
* Have an active or history of autoimmune disease or immune deficiency
* Have a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis based on a screening chest computed tomography (CT) scan
* Active tuberculosis
* Severe infections within 4 weeks
* Have received therapeutic oral or IV antibiotic medication within 2 weeks, except prophylactic antibiotic medication
* Have significant cardiovascular disease
* Are administered treatment with a live attenuated vaccine within 4 weeks, or anticipation of need for such a vaccine during the course of the study
* Have prior allogeneic bone marrow transplantation or solid organ transplant
* History of treatment with systemic immunostimulatory agents (including but not limited to interferons, interleukin-2) within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to initiation of study treatment
* History of treatment with systemic immunosuppressive medications within 2 weeks except acute, low-dose, systemic immunosuppressant medications, corticosteroids for chronic obstructive pulmonary disease and asthma, or mineralocorticoids and low-dose corticosteroids for participants with orthostatic hypotension or adrenocortical insufficiency
* Have a history or clinical evidence of any untreated CNS disease, seizures not controlled with standard medical therapy, or history of cerebrovascular accident (stroke), transient ischemic attack or subarachnoid hemorrhage within 6 months

AFT-50A Specific Exclusion Criteria:

● Prior treatment with T-cell costimulating or immune checkpoint blockade therapies including, but not limited to, CD137 agonists, anti-PD-1, anti-PD-L1, and anti-CTLA-4 therapeutic antibodies

Note: Additional study cohort specific inclusion and exclusion criteria may apply based on cohort assignment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed overall response rate (ORR) of each biomarker cohort | 48 Months
  AFT-50A Protocol: Overall response rate for each biomarker cohort is defined as the proportion of participants achieving a complete (CR) or partial (PR) response on two consecutive occasions at least 4 weeks apart, as determined by the investigator from AFT50A Protocol: Tumor assessments per RECIST v1.1.
The proportion of participants in each biomarker cohort who remain alive and progression-free for at least 6 months | 6 Months
  AFT-50B Protocol: Progression free survival rate at 6 months is defined as the proportion of participants who have not experienced disease progression or death from any cause at 6 months, as determined by the investigator according to RECIST v1.1

SECONDARY OUTCOMES:
Relative proportion of participants in each biomarker cohort who remain progression-free for at least 6 months compared to that from historical control studies | 6 Months per cohort
  AFT-50A Protocol: PFS rate at 6 months is defined as the proportion of participants who have not experienced disease progression or death from any cause at 6 months, as determined by the investigator according to RECIST v1.1
Investigator assessed disease-control rate of each biomarker cohort | 48 Months
  AFT-50A Protocol: Disease-control rate is defined as the proportion of participants achieving either stable disease, complete response, or partial response.
Duration of response for participants in each biomarker cohort who achieve a complete or partial response. | 48 Months
  AFT-50A Protocol: Duration of response is defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Overall survival (OS) rates of participants in each biomarker cohort after 24 months | 24 Months per cohort
  AFT-50A Protocol: 24-month overall survival rate is defined as the proportion of participants who have not experienced death from any cause at 24 months.
Investigator assessed disease-control rate of each biomarker cohort | 48 Months
  AFT-50B Protocol: Disease control rate is defined as the proportion of participants achieving either stable disease, complete response, or partial response at any time.
Duration of response for participants in each biomarker cohort who achieve a confirmed response (complete or partial) | 48 Months
  AFT-50B Protocol: Duration of response is defined as the time from the first occurrence of a documented objective response (complete or partial) to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Overall survival rates of participants in each biomarker cohort | 24 Months
  AFT-50B Protocol: 24-month overall survival rate is defined as the proportion of participants who have not experienced death from any cause at 24 months.

OTHER OUTCOMES:
Safety of each biomarker cohort: adverse events | 48 Months
  AFT-50A Protocol: The incidence and severity of adverse events, with severity determined according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0), as well as summaries of changes in clinically relevant laboratory test results, changes in vital signs, and study treatment exposures for each biomarker cohort
The safety of each biomarker cohort: Adverse Events | 48 Months
  AFT-50B Protocol: The incidence and severity of adverse events, with severity determined according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0). Summaries of changes in clinically relevant laboratory test results, changes in vital signs, and study treatment exposures for each biomarker cohort
Assess exploratory biomarkers in tumor tissue and peripheral blood, and their association with other molecular characteristics, disease status and/or participant response to study treatment | 48 Months
  AFT-50A and AFT-50B Protocols: Association of exploratory biomarkers with clinical outcomes, including but not limited to molecular analysis of tumor tissue and peripheral blood, as well as cytokine/chemokine and cellular analysis of peripheral blood.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Medstar Georgetown Cancer Institute, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University of Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Maine Medical Center, Scarborough, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Englewood Health, Englewood, New Jersey
  - Atlantic Health Systems/Morristown Medical Center, Morristown, New Jersey
  - Roswell Park, Buffalo, New York
  - Weill Cornell Medicine, New York, New York
  - Duke University Cancer Center, Durham, North Carolina
  - University of Oklahoma Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Portland Cancer Institute, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lifespan - Rhode Island Hospital, Providence, Rhode Island
  - Baptist Memorial Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aghajanian C, Sill MW, Darcy KM, Greer B, McMeekin DS, Rose PG, Rotmensch J, Barnes MN, Hanjani P, Leslie KK. Phase II trial of bevacizumab in recurrent or persistent endometrial cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2011 Jun 1;29(16):2259-65. doi: 10.1200/JCO.2010.32.6397. Epub 2011 May 2. PMID 21537039
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Rous J, Rems J, Cermak Z. [Extraction of peripherally located bronchial foreign bodies using a x-ray picture amplifier with a television loop]. Cesk Otolaryngol. 1975 Dec;24(6):335-41. No abstract available. Czech. PMID 1204078
- [Background] Rosenberg JE, Hoffman-Censits J, Powles T, van der Heijden MS, Balar AV, Necchi A, Dawson N, O'Donnell PH, Balmanoukian A, Loriot Y, Srinivas S, Retz MM, Grivas P, Joseph RW, Galsky MD, Fleming MT, Petrylak DP, Perez-Gracia JL, Burris HA, Castellano D, Canil C, Bellmunt J, Bajorin D, Nickles D, Bourgon R, Frampton GM, Cui N, Mariathasan S, Abidoye O, Fine GD, Dreicer R. Atezolizumab in patients with locally advanced and metastatic urothelial carcinoma who have progressed following treatment with platinum-based chemotherapy: a single-arm, multicentre, phase 2 trial. Lancet. 2016 May 7;387(10031):1909-20. doi: 10.1016/S0140-6736(16)00561-4. Epub 2016 Mar 4. PMID 26952546
- [Background] Schwartz LH, Seymour L, Litiere S, Ford R, Gwyther S, Mandrekar S, Shankar L, Bogaerts J, Chen A, Dancey J, Hayes W, Hodi FS, Hoekstra OS, Huang EP, Lin N, Liu Y, Therasse P, Wolchok JD, de Vries E. RECIST 1.1 - Standardisation and disease-specific adaptations: Perspectives from the RECIST Working Group. Eur J Cancer. 2016 Jul;62:138-45. doi: 10.1016/j.ejca.2016.03.082. Epub 2016 May 26. PMID 27237360
- [Background] Rini BI, Powles T, Atkins MB, Escudier B, McDermott DF, Suarez C, Bracarda S, Stadler WM, Donskov F, Lee JL, Hawkins R, Ravaud A, Alekseev B, Staehler M, Uemura M, De Giorgi U, Mellado B, Porta C, Melichar B, Gurney H, Bedke J, Choueiri TK, Parnis F, Khaznadar T, Thobhani A, Li S, Piault-Louis E, Frantz G, Huseni M, Schiff C, Green MC, Motzer RJ; IMmotion151 Study Group. Atezolizumab plus bevacizumab versus sunitinib in patients with previously untreated metastatic renal cell carcinoma (IMmotion151): a multicentre, open-label, phase 3, randomised controlled trial. Lancet. 2019 Jun 15;393(10189):2404-2415. doi: 10.1016/S0140-6736(19)30723-8. Epub 2019 May 9. PMID 31079938
- [Background] Colle R, Cohen R, Cochereau D, Duval A, Lascols O, Lopez-Trabada D, Afchain P, Trouilloud I, Parc Y, Lefevre JH, Flejou JF, Svrcek M, Andre T. Immunotherapy and patients treated for cancer with microsatellite instability. Bull Cancer. 2017 Jan;104(1):42-51. doi: 10.1016/j.bulcan.2016.11.006. Epub 2016 Dec 13. PMID 27979364
- [Background] Westin SN, Sill MW, Coleman RL, Waggoner S, Moore KN, Mathews CA, Martin LP, Modesitt SC, Lee S, Ju Z, Mills GB, Schilder RJ, Fracasso PM, Birrer MJ, Aghajanian C. Safety lead-in of the MEK inhibitor trametinib in combination with GSK2141795, an AKT inhibitor, in patients with recurrent endometrial cancer: An NRG Oncology/GOG study. Gynecol Oncol. 2019 Dec;155(3):420-428. doi: 10.1016/j.ygyno.2019.09.024. Epub 2019 Oct 15. PMID 31623857
- [Background] LoRusso PM. Inhibition of the PI3K/AKT/mTOR Pathway in Solid Tumors. J Clin Oncol. 2016 Nov 1;34(31):3803-3815. doi: 10.1200/JCO.2014.59.0018. Epub 2016 Sep 30. PMID 27621407
- [Background] Correction: A First-in-Human Phase I Study of the ATP-Competitive AKT Inhibitor Ipatasertib Demonstrates Robust and Safe Targeting of AKT in Patients with Solid Tumors. Cancer Discov. 2018 Nov;8(11):1490. doi: 10.1158/2159-8290.CD-18-1114. No abstract available. PMID 30385525
- [Background] Xue G, Zippelius A, Wicki A, Mandala M, Tang F, Massi D, Hemmings BA. Integrated Akt/PKB signaling in immunomodulation and its potential role in cancer immunotherapy. J Natl Cancer Inst. 2015 Jun 11;107(7):djv171. doi: 10.1093/jnci/djv171. Print 2015 Jul. PMID 26071042
- [Background] Cancer Genome Atlas Research Network; Kandoth C, Schultz N, Cherniack AD, Akbani R, Liu Y, Shen H, Robertson AG, Pashtan I, Shen R, Benz CC, Yau C, Laird PW, Ding L, Zhang W, Mills GB, Kucherlapati R, Mardis ER, Levine DA. Integrated genomic characterization of endometrial carcinoma. Nature. 2013 May 2;497(7447):67-73. doi: 10.1038/nature12113. PMID 23636398
- [Background] Miyasaka A, Oda K, Ikeda Y, Wada-Hiraike O, Kashiyama T, Enomoto A, Hosoya N, Koso T, Fukuda T, Inaba K, Sone K, Uehara Y, Kurikawa R, Nagasaka K, Matsumoto Y, Arimoto T, Nakagawa S, Kuramoto H, Miyagawa K, Yano T, Kawana K, Osuga Y, Fujii T. Anti-tumor activity of olaparib, a poly (ADP-ribose) polymerase (PARP) inhibitor, in cultured endometrial carcinoma cells. BMC Cancer. 2014 Mar 13;14:179. doi: 10.1186/1471-2407-14-179. PMID 24625059
- [Background] Gockley AA, Kolin DL, Awtrey CS, Lindeman NI, Matulonis UA, Konstantinopoulos PA. Durable response in a woman with recurrent low-grade endometrioid endometrial cancer and a germline BRCA2 mutation treated with a PARP inhibitor. Gynecol Oncol. 2018 Aug;150(2):219-226. doi: 10.1016/j.ygyno.2018.05.028. Epub 2018 Jun 22. PMID 29937315
- [Background] Jiao S, Xia W, Yamaguchi H, Wei Y, Chen MK, Hsu JM, Hsu JL, Yu WH, Du Y, Lee HH, Li CW, Chou CK, Lim SO, Chang SS, Litton J, Arun B, Hortobagyi GN, Hung MC. PARP Inhibitor Upregulates PD-L1 Expression and Enhances Cancer-Associated Immunosuppression. Clin Cancer Res. 2017 Jul 15;23(14):3711-3720. doi: 10.1158/1078-0432.CCR-16-3215. Epub 2017 Feb 6. PMID 28167507
- [Background] Strickland KC, Howitt BE, Shukla SA, Rodig S, Ritterhouse LL, Liu JF, Garber JE, Chowdhury D, Wu CJ, D'Andrea AD, Matulonis UA, Konstantinopoulos PA. Association and prognostic significance of BRCA1/2-mutation status with neoantigen load, number of tumor-infiltrating lymphocytes and expression of PD-1/PD-L1 in high grade serous ovarian cancer. Oncotarget. 2016 Mar 22;7(12):13587-98. doi: 10.18632/oncotarget.7277. PMID 26871470
- See also: CTCAE Version 5.0 — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm